CLINICAL TRIAL: NCT05092711
Title: Cardiovascular Risk Factors , Complications and Threputic Management Strategies in Patients With Coronary Heart Disease and COVID 19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Marghany Hassan Mohamed, Ahmed Marghany Hassan Mohammed, Assiut University
Other Study IDs: COVIHD
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- in patients with coronary heart disease and COVID 19
  Interventions: Behavioral: Observation; Drug: Observation

INTERVENTIONS:
Behavioral: Observation — Using INTERASPIRE model to determine patients with established CHD whether the guidelines on cardiovascular disease prevention are being followed or not with incorporation of COVID 19 as a risk factor with the other classical risk factors to understand significance of the new pandemic virus in mortality and morbidity of CVD and coronary events in association with the other known classical risk factors .
Drug: Observation — Using INTERASPIRE model to determine patients with established CHD whether the guidelines on cardiovascular disease prevention are being followed or not with incorporation of COVID 19 as a risk factor with the other classical risk factors to understand significance of the new pandemic virus in mortality and morbidity of CVD and coronary events in association with the other known classical risk factors .

SUMMARY:
Using INTERASPIRE model to determine patients with established CHD whether the guidelines on cardiovascular disease prevention are being followed or not with incorporation of COVID 19 as a risk factor with the other classical risk factors to understand significance of the new pandemic virus in mortality and morbidity of CVD and coronary events in association with the other known classical risk factors .

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a class of diseases that involve the heart or blood vessels, CVD includes coronary artery diseases (CAD) such as angina and myocardial infarction (commonly known as a heart attack. Other CVDs include stroke, heart failure, hypertensive heart disease, rheumatic heart disease, cardiomyopathy, abnormal heart rhythms, congenital heart disease, valvular heart disease, carditis, aortic aneurysms, peripheral artery disease, thromboembolic disease, and venous thrombosis.

At the 65th World Health Assembly in May 2012 Ministers of Health and Senior Health Officials from the 194 WHO member states adopted a global target to reduce premature mortality from non-communicable diseases (NCDs), and in particular cardiovascular disease, by 25% by 2025. The main objectives of CVD prevention are to reduce cardiovascular morbidity and mortality, improve quality of life, and increase life expectancy.

The 52 country INTERHEART study has shown that the classical risk factors for CHD account for most of the risk of myocardial infarction worldwide. This scientific evidence has led to international, regional and national guidelines on CVD prevention, which define patient priorities for preventive action and lifestyle and treatment goals

1. In 1994, 1998, 2003, 2007, 2012 and 2016. [3-7]. The European Society of Cardiology together with other partner Societies has engaged in a comprehensive programme of CVD prevention in clinical practice since 1994 with the acronym EUROASPIRE (European Action on Secondary and Primary Prevention by Intervention to Reduce Events)
2. in 2012: Ministers of Health and Senior Health Officials: adopted a global target to reduce premature mortality from non-communicable diseases (NCDs), and in particular cardiovascular disease, by 25% by 2025.
3. In [2], 2013 : The 52 country INTERHEART study has shown that the classical risk factors for CHD account for most of the risk of myocardial infarction worldwide.

The INTERASPIRE survey began when the ESC Euro Observational Research Programme decided to expand the EUROASPIRE programme to include other WHO regions, starting with a pilot study in Malaysia and Argentina in 2019. The main survey (2020-2022) is now being organised in partnership with the World Heart Federation, Asia Pacific Society of Cardiology, InterAmerican Society of Cardiology and the Pan-African Society of Cardiology and includes selected countries in all 6 WHO regions: African Region, Region of Americas, Eastern Mediterranean Region, European Region, South-East Asia Region, and Western Pacific Region.

* This international study is being conducted through National Societies of Cardiology which have responsibility for appointing National Coordinators, selecting geographical regions (minimum of three) and hospital centres (minimum of 6 in each country) together with Principal Investigators.
* The study population is a consecutive sample of coronary patients from each hospital which meet the following diagnostic criteria: Acute coronary syndromes (acute myocardial infarction with ST elevation (STEMI) and Non ST elevation MI (Non-STEMI) and stable coronary artery disease). Patients are interviewed and examined in hospital using standardised methodology, including one central laboratory in Helsinki, Finland, for measurement of fasting lipids, glucose, HbA1c, creatinine and urinary albumin, and then followed up for hospitalisations, non-fatal and fatal cardiovascular events and all cause mortality.

Using INTERASPIRE model to determine patients with established CHD whether the guidelines on cardiovascular disease prevention are being followed or not with incorporation of COVID 19 as a risk factor with the other classical risk factors to understand significance of the new pandemic virus in mortality and morbidity of CVD and coronary events in association with the other known classical risk factors .

ELIGIBILITY:
Inclusion Criteria:

150 consecutive patients, men or women [≥18 years and <80 years at the time of identification]

* Patient s may fulfil more than one of the following diagnostic criteria:
* Elective CABG.
* Elective PCI.
* Acute coronary syndromes (acute myocardial infarction with ST elevation (STEMI) and Non ST elevation MI (Non-STEMI) including those treated with primary PCI and/or CABG, and unstable angina).

It is recognised that hospital diagnoses for AMI, and unstable angina without evidence of infarction, may not always meet the World Heart Organisation (WHO) or other standard diagnostic criteria. However, it is important to include all cases diagnosed as AMI or unstable angina in hospital clinical practice because, as a consequence of these diagnoses, they should all have received appropriate management for secondary prevention.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: will be taken as 150 patients from patients attending Assiut University Heart Hospital outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
• To determine in patients with established CHD (acute myocardial infarction and ischaemia and patients following revascularisation by angioplasty or coronary artery surgery) whether the guidelines on cardiovascular disease prevention are being followed. | 1.5 year
• To follow-up all patients one year after the interview for hospitalisations, cardiovascular procedures, cardiovascular events and cardiovascular and all cause mortality | 1.5 year
• To describe the prevalence of cardiovascular risk factors, acute and long-term cardiovascular complications and therapeutic management in patients with CHD and COVID-19 | 1.5 year
• To compare the risk factor profiles in CHD patients with and without a history of COVID-19 | 1.5 year
• To compare the diagnostic and therapeutic strategies in CHD patients with and without a history of COVID-19 | 1.5 year
• To compare the acute and long-term cardiovascular complications in CHD patients with and without a history of COVID-19 | 1.5 year

SECONDARY OUTCOMES:
• To compare diagnostic and therapeutic strategies in prevalent cases of familial hypercholesterolaemia in patients with established coronary disease and the residual risk among these patients with current treatments. | 1.5 year
• To compare diagnostic and therapeutic strategies in patients with established coronary disease in relation to glucose metabolism (impaired fasting glycaemia, impaired glucose tolerance and diabetes). | 1.5 year
• To follow-up all patients one year after the interview for hospitalisations, cardiovascular procedures, cardiovascular events and cardiovascular and all cause mortality | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AboelKasem farghal, Professor, Study Director — Assiut University; Hossam Hassan Ali Elaraby, Professor, Study Director — Assiut University
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided